CLINICAL TRIAL: NCT04593342
Title: Evaluation of the Efficacy of B-Cure Laser Treatment on Pain and Functionality Following Arthroscopic Rotator Cuff Repair: A Prospective Double Blind, Randomized, Sham-Controlled Clinical Study
Brief Title: Photobiomodulation Laser Therapy Following Arthroscopic Rotator Cuff Repair
Acronym: LLL&RotC01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erika Carmel ltd (Other)
Collaborators: Holy Family Hospital, Methuen, MA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HFH-219-2020
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Rotator Cuff Tears
Keywords: Photobiomodulation; Low-Level Laser Therapy
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Single center, Prospective, Double Blind, Randomized, Sham-Controlled, Parallel Group, Superiority comparison
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard + B-Cure Pro (Active Comparator): Subjects from the Standard + B-Cure Pro group will receive standard care and in addition will self-treat at home with the B-Cure device
  Interventions: Device: B-Cure Pro
- Standard + Sham (Sham Comparator): Subjects from the Standard + Sham group will receive standard care and in addition will self-treat at home with the sham B-Cure device
  Interventions: Device: Sham

INTERVENTIONS:
Device: B-Cure Pro — The B-Cure laser Pro is a portal, non-invasive, low level laser therapy device, that emits light in the near infrared (808nm) over an area of 1X4.5 cm2 with power output of 250mW, and energy dose of 5J/min.
  Arms: Standard + B-Cure Pro
Device: Sham — The sham device is externally identical to the B-Cure Pro and emit the same guiding light, but does not emit the therapeutic near infrared rays.
  Arms: Standard + Sham

SUMMARY:
Rehabilitation following rotator cuff surgery is characterized with high levels of pain, limited range of motion, and decreased quality of life. The purpose of this study is to evaluate the B-Cure laser photobiomodulation home-use device in addition to standard care, for the reduction of pain, increase in functionality, and improvement of life quality during rehabilitation following rotator cuff arthroscopic surgery.

DETAILED DESCRIPTION:
Patients planned to undergo rotator cuff arthroscopy will be randomized to receive active or sham devices for self-application at home in addition to standard care. Patients will be invited to up to 5 visits at the clinic: baseline (before surgery), post-operative day 1, and 1, 3, and optionally 6 months after surgery. Evaluations will include physical examination, physical activity tests, range of motion measurements, Constant score, thermal imaging, and patient reported outcomes including subjective pain level by visual analogue scale, functional and quality of life questionnaires.

The study hypothesis is that B-Cure laser treatments, applied, at home, by the patient, can reduce pain and accelerate healing over standard care thereby improving the rehabilitation process following rotator cuff arthroscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65
* Men or women
* Full or partial rotator cuff tear
* Scheduled to undergo RCAS because of failure of conservative therapy (injections, medication, physiotherapy)
* Is willing to perform the full protocol
* Voluntarily sign and date an informed consent form
* Be able to understand and complete the various questionnaires

Exclusion Criteria:

* Is unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits
* Participation in another clinical study within 30 days before screening
* Scheduled to undergo an elective medical procedure during the study timeframe that will interfere with the study as deemed by the PI
* Pregnant
* Has any photobiomodulation (low level laser) device at home or has previously used photobiomodulation for shoulder pain
* Use of medications, herbal supplements, perfumes or cosmetics that may affect sensitivity to light
* Has osteoarthritis
* Other chronic pain conditions: fibromyalgia, failed back surgery, back pain
* Avascular necrosis
* Rheumatoid arthritis
* Psychiatric disorders including major depression, schizophrenia, bipolar disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in level of pain by VAS | 1 month post-surgery
  Subject assessment of pain will be evaluated using a Visual Analogue Scale (VAS), were 0 is "no pain" and 100 is "intolerable pain".

SECONDARY OUTCOMES:
Change from baseline in functionality (CONSTANT score) | 1 month post-surgery
  The CONSTANT score used to assess the functionality of the shoulder by clinicians. The range of the score is 0-100. The higher the score, the higher the quality of the function.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Hadad, MD, Principal Investigator — Department of Orthopedic Surgery, Holy Family Hospital, Nazareth
Locations (1):
- Holy Family Hospital, Nazareth, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abufoul R, Gavish L, Haddad M. Photobiomodulation self-treatment at home after rotator cuff arthroscopic repair accelerates improvement in pain, functionality, and quality of life: A double-blind, sham-controlled, randomized clinical trial. Lasers Surg Med. 2023 Sep;55(7):662-673. doi: 10.1002/lsm.23692. Epub 2023 Jun 8. PMID 37288499